CLINICAL TRIAL: NCT07315087
Title: A Clinical Study Evaluating the Safety and Preliminary Efficacy of Universal Allogeneic CAR T-cell Therapy Targeting CD19 and BCMA(QT-019C) in Patients With Relapse/Refractory Autoimmune Diseases
Brief Title: CAR T-cell Therapy Targeting CD19 and BCMA(QT-019C) in Patients With Relapse/Refractory Autoimmune Diseases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Shanghai Xiniao Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025138
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: SLE - Systemic Lupus Erythematosus; SSc-Systemic Sclerosis; IIM- Idiopathic Inflammatory Myopathies; ANCA Associated Vasculitis (AAV); Connective Tissue Disease-Associated Thrombocytopenia; SLE-ITP
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QT-019C (Experimental): Universal allogeneic anti-CD19/BCMA CAR T-cells. Biological/Vaccine: universal allogeneic anti-CD19/BCMA
  Interventions: Biological: QT-019C

INTERVENTIONS:
Biological: QT-019C — universal allogeneic anti-CD19/BCMA CAR T-cells

SUMMARY:
CAR T-cell Therapy Targeting CD19 and BCMA(QT-019C) in Patients With Relapse/Refractory Autoimmune Diseases

DETAILED DESCRIPTION:
This is an investigator-initiated trial to evaluate the safety and efficacy of universal allogeneic anti-CD19/BCMA CAR T-cells(QT-019C) in Patients With Relapse/Refractory Autoimmune Diseases.Study intervention consists of a single infusion of universal allogeneic CART-cells administered intravenously after a lymphodepleting therapy regimen of cyclophosphamide.Interim analysis will be performed when participants finish the visit at 12 and 24 weeks after CAR T-cell infusion.

ELIGIBILITY:
Inclusion Criteria:

Common Inclusion Criteria:

1. Age ≥ 18 years old (inclusive), regardless of gender.
2. Functional requirements for major organs are as follows（Except for abnormalities related to autoimmune disease activity）: 1) Bone marrow function must meet: A. Neutrophil count ≥ 1×109/L (no colony-stimulating factor treatment within 2 weeks before examination); B. Hemoglobin ≥ 60g/L; 2) Liver function: Alanine aminotransferase (ALT) ≤ 3×ULN (excluding ALT elevation due to inflammatory myopathy), aspartate aminotransferase (AST)≤3×Upper limit of normal (ULN) (excluding AST elevation due to inflammatory myopathy), TBIL≤2×ULN (or ≤ 3.0×ULN for subjects with Gilbert syndrome); 3) Renal function: creatinine clearance rate (CrCl) ≥ 30mL/minute (calculated by Cockcroft/Gault formula, acute CrCl decrease due to the target disease is excluded; LN is excluded).
3. Female subjects of childbearing potential and male subjects with partners of childbearing potential must use medically approved contraception or abstinence during the study treatment period and for at least 6 months after the end of the study treatment; Female subjects of childbearing potential must have a negative human chorionic gonadotropin (hCG) test within 7 days before study enrollment and not be lactating.
4. Willing to participate in this clinical study, sign an informed consent form, have good compliance, and cooperate with follow-up.

Disease-Specific Inclusion Criteria:

Refractory/Relapsed Systemic Lupus Erythematosus:

1. SLE meeting the 2019 American College of Rheumatology (ACR) /European League Against Rheumatism (EULAR) and classification criteria.
2. Disease activity score SLEDAI-2000 ≥ 8; or with significant organ involvement, such as lupus nephritis (histologically confirmed active nephritis of class III or IV, with or without class V, with an NIH activity index > 2, evidence of increased chronicity index; urine protein-to-creatinine ratio > 1.0 g/g, or 24-hour urinary protein > 1.0 g).
3. Definition of refractory or relapsing disease: lack of response after more than 6 months of conventional therapy, or recurrence of disease activity after remission. Conventional therapy is defined as treatment with glucocorticoids in combination with one or more of the following immunomodulatory agents: cyclophosphamide, antimalarial drugs, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, as well as biologics such as rituximab, belimumab, and telitacicept.

Refractory/Relapsed/Progressive Systemic Sclerosis:

1. Scleroderma fulfilling the 2013 ACR classification criteria.
2. Positive scleroderma-related antibodies.
3. Presence of diffuse cutaneous sclerosis or active interstitial lung disease (high-resolution computed tomography (HRCT) showing ground-glass opacities).
4. Definition of relapsed/refractory: Conventional treatment over 6 months remains ineffective, or disease recurrence after remission. Definition of conventional treatment: the use of glucocorticoids , and any one or more of the following immunomodulatory drugs: cyclophosphamide, antimalarials, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, and biologics including belimumab, rituximab, and tocilizumab, etc.
5. Definition of progressive: Rapid skin progression (mRSS increase > 25%); or progression of lung disease (forced vital capacity (FVC) decrease by 10%, or FVC decrease by more than 5% with diffusing capacity of the lung for carbon monoxide (DLCO) decrease by 15%).

Note: Meeting either criterion 4 or 5 is sufficient.

Refractory/Relapsed/Progressive Inflammatory Myopathy:

1. Inflammatory myopathy fulfilling the 2017 EULAR/ACR classification criteria (including Dermatomyositis (DM), Polymyositis (PM), Anti-Synthetase Syndrome (ASS), and Necrotizing Myopathy (NM)).
2. Muscle involvement with Manual Muscle Testing-8 (MMT-8) score less than 142 and at least two abnormalities found among the following five core measurements (Physician Global Assessment (PhGA), Patient Global Assessment (PtGA), or extramuscular disease activity score ≥ 2; Health Assessment Questionnaire (HAQ) total score ≥ 0.25; muscle enzyme levels ≥ 1.5×ULN);
3. Definition of relapsed/refractory: Conventional treatment over 6 months remains ineffective, or disease recurrence after remission. Definition of conventional treatment: the use of glucocorticoids , and any one or more of the following immunomodulatory drugs: cyclophosphamide, antimalarials, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, and biologics including belimumab, rituximab, and tocilizumab, etc.
4. Definition of progressive: Rapid progression of interstitial lung disease within a short period.

Note: Meeting either criterion 3 or 4 is sufficient.

Refractory/Relapsed ANCA-Associated Vasculitis:

1. ANCA-Associated Vasculitis fulfilling 2022 ACR/EULAR criteria, including microscopic polyangiitis, granulomatosis with polyangiitis, and eosinophilic granulomatosis with polyangiitis.
2. Positive ANCA-associated antibodies (MPO-ANCA or PR3-ANCA positive).
3. The Birmingham Vasculitis Activity Scale (BVAS) ≥ 15 points (a total score of 63 points), indicating active vasculitis.
4. Definition of refractory/relapsed: Conventional treatment over 6 months remains ineffective, or disease recurrence after remission., or disease recurrence after remission. Definition of conventional treatment: the use of glucocorticoids and any one or more of the following immunomodulatory drugs: cyclophosphamide, antimalarials, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, and biologics including belimumab, rituximab, and tocilizumab, etc.

Refractory/Relapsed Connective Tissue Disease-associated thrombocytopenia:

1. Diagnosis of connective tissue disease established according to the latest classification criteria, including but not limited to systemic lupus erythematosus, primary Sjögren's syndrome, antiphospholipid syndrome, and undifferentiated connective tissue disease.
2. Confirmed diagnosis of connective tissue disease-associated thrombocytopenia, with platelet count <30 × 10^9/L, or <50 × 10^9/L accompanied by a bleeding tendency.
3. Bone marrow morphology consistent with immune thrombocytopenia.
4. Prior treatment with at least one course of corticosteroid pulse therapy, or high-dose corticosteroids in combination with one or more immunosuppressants (including biologics) for at least 3 months, without achieving partial remission, or inability to maintain efficacy during steroid tapering.

Exclusion Criteria:

1. Subjects with a history of severe drug allergies or allergic tendencies.
2. Presence or suspicion of uncontrolled or treatment-required fungal, bacterial, viral, or other infections.
3. Subjects with central nervous system diseases caused by autoimmune diseases or non-autoimmune diseases (including epilepsy, psychosis, organic brain syndrome, cerebral vascular accidents, encephalitis, central nervous system vasculitis).
4. Subjects with insufficient cardiac function.
5. Subjects with congenital immunoglobulin deficiencies.
6. History of malignancy within five years.
7. Subjects with end-stage renal failure(LN is excluded).
8. Subjects who are positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with peripheral blood HBV DNA >ULN; subjects positive for hepatitis C virus (HCV) antibody and peripheral blood HCV RNA; individuals positive for human immunodeficiency virus (HIV) antibody; individuals positive for syphilis testing.
9. Subjects with psychiatric disorders and severe cognitive impairments.
10. Subjects who have participated in other clinical trials within the past 3 months prior to enrollment.
11. Subjects who have received immunosuppressive agents or biologics with therapeutic effects for indications within 5 half-life prior to enrollment.
12. Pregnant women or women planning to conceive.
13. Subjects whom the investigator believes have other reasons that make them unsuitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-18 (Estimated)

PRIMARY OUTCOMES:
The number and severity of dose-limiting toxicity (DLT) events | Within 28 Days After QT-019C infusion
  DLT will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, and the ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells.
The total number, incidence, and severity of AEs | Up to 12 Months After QT-019C Infusion
  2. The total number, incidence, and severity of AEs

SECONDARY OUTCOMES:
Clinical response of R/R AIDs | Up to 24 Months After UCAR T-cell Infusion
  Clinical response of R/R AIDs

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No